CLINICAL TRIAL: NCT02980874
Title: SAPPHIRE: A Randomized, Masked, Controlled Trial To Study The Safety And Efficacy Of Suprachoroidal CLS-TA In Conjunction With Intravitreal Aflibercept In Subjects With Retinal Vein Occlusion
Brief Title: Suprachoroidal Injection of Triamcinolone Acetonide With IVT Aflibercept in Subjects With Macular Edema Following RVO
Acronym: SAPPHIRE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Primary, 8-week efficacy endpoint not achieved. No additional benefit for subjects receiving a corticosteroid together with an intravitreal anti-VEGF agent.
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLS1003-301
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Macular Edema; Retinal Vein Occlusion
Keywords: RVO; ME; Central Subfield Thickness; OCT; Optical Coherence Tomography; Cystoid Macular Edema; Subretinal Fluid; Eylea; Aflibercept; Anti-VEGF; Suprachoroidal; Triamcinolone acetonide
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Triamcinolone Acetonide; aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): IVT aflibercept (2 mg/0.05 mL) + CLS-TA (4 mg/100 µL) SC injections
  Interventions: Drug: suprachoroidal CLS-TA; Drug: IVT aflibercept
- Control (Active Comparator): IVT aflibercept (2 mg/0.05 mL) + sham SC procedure
  Interventions: Drug: suprachoroidal sham; Drug: IVT aflibercept

INTERVENTIONS:
Drug: suprachoroidal CLS-TA — suprachoroidal injection of CLS-TA
  Other Names: Triamcinolone acetonide
  Arms: Active
Drug: suprachoroidal sham — suprachoroidal sham procedure
  Arms: Control
Drug: IVT aflibercept — 2 mg intravitreal injection of aflibercept
  Other Names: Aflibercept

SUMMARY:
This is a Phase 3, multicenter, randomized, masked, controlled, parallel group study of 12 months duration in treatment naïve subjects with RVO.

DETAILED DESCRIPTION:
A randomized, masked, controlled trial to study the safety and efficacy of suprachoroidal CLS-TA in conjunction with intravitreal aflibercept in subjects with retinal vein occlusion

ELIGIBILITY:
Inclusion Criteria:

* Has a clinical diagnosis of RVO in the study eye
* Has a CST of ≥ 300 µm in the study eye
* Has an ETDRS BCVA score of ≥ 20 letters read and ≤ 70 letters read in the study eye;
* Is naïve to local pharmacologic treatment for RVO in the study eye;

Exclusion Criteria:

* Any active ocular disease or infection in the study eye other than RVO
* History of glaucoma, intraocular pressure > 21 mmHg or ocular hypertension requiring more than one medication
* Any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study
* Any evidence of neovascularization in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ciulla, MD MBA, Study Director — Clearside Biomedical, Inc.
Locations (110):
- United States (58):
  - Associated Retina Consultants, Ltd., Peoria, Arizona
  - Retinal Consultants of Arizona and Retinal Research Institute, Phoenix, Arizona
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Associated Retina Consultants, Ltd., Phoenix, Arizona
  - Retina Centers P.C., Tucson, Arizona
  - California Retina Research Consultants, Bakersfield, California
  - Retina Vitreous Medical Group Clinical Research, Beverly Hills, California
  - Atlantis Eyecare, Huntington Beach, California
  - Jacobs Retina Center at the Shiley Eye Institute, UCSD, La Jolla, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - East Bay Retina Consultants Inc., Oakland, California
  - Southern California Desert Retina Consultants, Palm Desert, California
  - Retina Institute of California, Palm Desert, California
  - Retina Consultants San Diego, Poway, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants CRC, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Colorado Retina Associates, Golden, Colorado
  - New England Retina Associates, Hamden, Connecticut
  - MedEye Associates, Miami, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Southeast Retina Center, PC, Augusta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - Illinois Eye and Ear Infirmary, UIC, Chicago, Illinois
  - Illinois Retina Associates, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Retina Associates, PA, Shawnee Mission, Kansas
  - Retina and Vitrous Associates of Kentucky, Lexington, Kentucky
  - Wilmer Eye Institute John Hopkins University, Baltimore, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - The Retina Institute, St Louis, Missouri
  - Retina Associates of NJ, Teaneck, New Jersey
  - Western Carolina Retinal Associates, PA, Asheville, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Cleveland Clinic Foundation/Cole Eye Institute, Cleveland, Ohio
  - Oregon Retina Institute, Medford, Oregon
  - Casey Eye Institute/Oregon Health & Science University, Portland, Oregon
  - Eye Care Specialists, Kingston, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates-Arlington, Arlington, Texas
  - Austin Retina Associates, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Valley Retina Institute, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - University of Utah HSC - John A. Moran Eye Center, Salt Lake City, Utah
  - Retina Institute of Virginia, Richmond, Virginia
  - Virginia Retina Center, Warrenton, Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin
- Australia (6):
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Save Site Institute, University of Sydney, Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Marsden Eye Specialists, Sydney, New South Wales
  - The Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria
  - Specialist Eye Group, Melbourne, Victoria
- Austria (2):
  - University of Graz-Department of Ophthalmology, Graz
  - Kepler University Hospital, Linz
- Canada (5):
  - UBC/VGH Eye Care Centre, Vancouver, British Columbia
  - St. Joseph's Health Care London, Ivey Eye Institute, London, Ontario
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - Institut de l'oeil des Laurentides, Boisbriand, Quebec
  - CIUSSS de l'Est-de-l'Ile-de-Montreal. Hospital Maisonneuve-Rosemont, Comite d'ethique de la recherche, Montreal, Quebec
- Denmark (2):
  - Rigshospitalet, Glostrup Municipality
  - Dept. of Ophthalmology, Sjællands Universitetshospital, Roskilde, Roskilde
- Hungary (6):
  - Semmelweis Egyetem, Szemeszeti Klinika, Budapest
  - Bajcsy-Zsilinszky Korhaz es Rendelointezet, Szemeszeti Osztaly, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Budapest Retina Associates, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Szemklinika, Debrecen
  - Ganglion Orvosi Kozpont, Pécs
- India (6):
  - M&J Western Regional Institute of Ophthalmology, Ahmedabad, Gujarat
  - T.N. Medical College and B.Y.L. Nair Charitable Hospital, Mumbai, Maharashtra
  - Department of Medical Ophthalmology, Retina & Uvea, Delhi, New Delhi
  - Aravind Eye Hospitals & Postgraduate Institute of Ophthalmology, Madurai, Tamil Nadu
  - Smt. Kanuri Santhamma Centre for Vitreo Retinal Diseases, Hyderabad, Telangana
  - Disha Eye Hospital Private Limited, Kolkata, West Bengal
- Bnai Zion Medical Center, Haifa, Israel
- ASST Fatebenefratelli Sacco - P.O.L., University of Milan, Dep. of Ophthalmology, Milan, Italy
- Philippines (3):
  - Cebu Doctor's University Hospital, Cebu City
  - Peregrine Eye & Laser Institute, Makati City
  - The Medical City, Pasig
- Poland (4):
  - Oftalmika sp. z o. o., Bydgoszcz
  - Optimum Profesorskie Centrum Okulistyki, Gdansk
  - Uniwersytet Medyczny w Lublinie, Lublin
  - Centrum Diagnostyki i Mikrochirurgii Oka Lens, Olsztyn
- Portugal (3):
  - Centro Clinico Academico Braga - 2CA-Braga, Braga
  - Centro Hospitalar e Universitario de Coimbra, E.P.E., Coimbra
  - Centro Hospitalar de Sao Joao, E.P.E., Porto
- Fakultna nemocnica s poliklinikou Zilina, Žilina, Slovakia
- Spain (8):
  - Instituto Cinico Quirurgico de Oftalmologia, Bilbao, Vizcaya
  - Hospital General de Catalunya, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Instituto Oftalmologico Fernandez-Vega, Oviedo
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Miguel Servet, Zaragoza
  - Hospital Clinico Universitario, Zaragoza
- Taiwan (2):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (2):
  - Queens University Royal Victoria Hospital Trust, Belfast
  - Sunderland Eye Infirmary, Sunderland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Control
Started | 231 | 229
Completed | 128 | 127
Not Completed | 103 | 102
Not completed — Adverse Event | 2 | 7
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Lost to Follow-up | 5 | 5
Not completed — Includes premature discontinuation due to study termination. | 88 | 88
Not completed — Unknown study completion status | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population included all randomly assigned subjects who were administered at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 231 | 229 | 460
Age, Categorical [Count of Participants; unit: Participants] — Age of patients in years relative to the date of the Screening visit.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 89 | 107 | 196
    >=65 years | 142 | 122 | 264
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age of patients in years relative to the date of the Screening visit.
  Years | 66.4 (12.31) | 64.9 (12.42) | 65.7 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 105 | 202
  Male | 134 | 124 | 258
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 33 | 40 | 73
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 12 | 22
  White | 181 | 177 | 358
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 6 | 1 | 7
  United States | 182 | 183 | 365
  Philippines | 0 | 3 | 3
  United Kingdom | 4 | 2 | 6
  Portugal | 3 | 2 | 5
  India | 13 | 19 | 32
  Spain | 3 | 2 | 5
  Canada | 2 | 3 | 5
  Taiwan | 2 | 1 | 3
  Denmark | 2 | 1 | 3
  Poland | 5 | 5 | 10
  Slovakia | 0 | 1 | 1
  Australia | 9 | 6 | 15
Type of Retinal Vein Occlusion [Count of Participants; unit: Participants]
  Branch retinal vein occlusion | 124 | 124 | 248
  Central retinal vein occlusion | 107 | 105 | 212

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Demonstrating ≥ 15 Letter Improvement From Baseline in Early Treatment of Diabetic Retinopathy Study (ETDRS)
Description: Best corrected visual acuity (BCVA) refers to the measurement of the best possible vision that can be achieved following refraction or correction. BCVA was assessed following the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol and was measured in the number of letters read correctly on an ETDRS eye chart. An increase from the pre-treatment state in BCVA of 15 letters or more represents a clinically meaningful improvement.
Time Frame: 2 months
Population: The Intent-to-treat population included all randomized subjects who received at least one study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Control
Number analyzed (Participants) | 231 | 229
Participants | 114 | 127
Statistical Analysis 1: Comparison: Active vs Control; Based on a Pearson chi-square test, a total sample size of approximately 460 subjects provided 90% power to detect a difference of 15% between the Active and Control arms assuming the Control arm showed a proportion of 0.50 at 8 weeks. The primary analysis was a test of superiority of the Active arm over the Control arm, and was based on a Cochran-Mantel-Haenszel chi-square test stratified by type of retinal vein occlusion; Test type: Superiority; p = 0.187, Cochran-Mantel-Haenszel — The a priori threshold for statistical significance was 0.050. Prior to evaluating the results of the CMH test, a Breslow-Day test with Tarone's adjustment was conducted to confirm the homogeneity of the odds ratios between RVO strata; The CMH test was stratified by the type of retinal vein occlusion, i.e., branch vs. central; Difference in percentages = -6.1, 95% CI 2-sided [-15.2 to 3.0] — Estimated value was calculated as the percentage of subjects in the Active arm meeting the primary endpoint minus the percentage of subjects in the Control arm meeting the primary endpoint

2. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity
Description: Best corrected visual acuity (BCVA) refers to the measurement of the best possible vision that can be achieved following refraction or correction. BCVA was assessed following the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol and was measured in the number of letters read correctly on an ETDRS eye chart. A positive change from baseline value represents an improvement in vision.
Time Frame: 6 months
Population: The Intent-to-treat population included all randomized subjects who received at least one study treatment.
Measure: Least Squares Mean (Standard Error); unit: Letters
Arm/Group | Active | Control
Number analyzed (Participants) | 231 | 229
Letters | 15.5 (0.85) | 20.5 (0.85)

3. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness
Description: Central subfield thickness (CST) is a diagnostic measurement used in identifying the presence of edema in the circular area 1 mm in diameter centered around the fovea. CST was measured using spectral domain optical coherence tomography (SD-OCT). A masked reading center graded the SD-OCT digital images. A negative change from baseline value represents a reduction in macular edema.
Time Frame: 6 months
Population: The Intent-to-treat population included all randomized subjects who received at least one study treatment.
Measure: Least Squares Mean (Standard Error); unit: Microns
Arm/Group | Active | Control
Number analyzed (Participants) | 231 | 210
Microns | -354.3 (8.01) | -416.2 (8.05)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 48 weeks of follow-up.
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 0/231 | 0/229
Serious Adverse Events (participants affected / at risk) | 25/231 | 28/229
Other Adverse Events (participants affected / at risk) | 128/231 | 83/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=231) | Control (N=229)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 0 (0) — #Fellow eye
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Visual acuity reduced (Eye disorders) | 2 (2) | 0 (0) — #Study eye
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) — #Study eye
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abasia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1) — #Study eye
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 3 (3) | 0 (0) — #Study eye
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rotor cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Paraganglion neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 3 (3)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=231) | Control (N=229)
Cataract (Eye disorders) | 21 (29) | 9 (12)
Cataract subcapsular (Eye disorders) | 20 (22) | 3 (3)
Conjunctival haemorrhage (Eye disorders) | 42 (65) | 28 (31)
Eye pain (Eye disorders) | 20 (24) | 11 (11)
Macular oedema (Eye disorders) | 8 (11) | 13 (16)
Visual acuity reduced (Eye disorders) | 16 (18) | 6 (7)
Vitreous detachment (Eye disorders) | 13 (16) | 9 (10)
Intraocular pressure increased (Investigations) | 33 (51) | 9 (13)
Nasopharyngitis (Infections and infestations) | 9 (9) | 13 (13)
Hypertension (Vascular disorders) | 15 (18) | 15 (17)

LIMITATIONS AND CAVEATS:
Due to the early termination of the trial by sponsor all planned study visits were not completed by all treated subjects; therefore, all planned data was not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institutions and Investigators participating in this study shall have no right to publish or present the results of this study without the prior written consent of Clearside Biomedical, Inc.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT02980874/Prot_SAP_000.pdf